CLINICAL TRIAL: NCT05712694
Title: ADI-PEG 20 or Placebo Plus Gemcitabine and Docetaxel in Previously Treated Subjects With Leiomyosarcoma (ARGSARC): A Randomized, Double Blind, Multi-Center Phase 3 Trial
Brief Title: Study of ADI-PEG 20 or Placebo Plus Gem and Doc in Previously Treated Subjects With Leiomyosarcoma (ARGSARC)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Polaris Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: POLARIS2022-001
Record Dates: First submitted 2022-12-13; First posted 2023-02-03 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Soft Tissue Sarcoma
Keywords: Soft Tissue Sarcoma; Arginine; Arginine Deiminase; ADI-PEG 20; Pegargiminase; Leiomyosarcoma
MeSH Terms: conditions — Sarcoma; Leiomyosarcoma | interventions — ADI PEG20

STUDY DESIGN:
Intervention Model Description: This is a global, multicenter, randomized, double-blind, placebo-controlled, parallel-group phase 3 trial that will compare the efficacy and safety in subjects with advanced or metastatic LMS previously treated with an anthracycline.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a global, multicenter, randomized, double-blind, placebo-controlled, parallel-group phase 3 trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ADIGemDoc (Experimental): ADI-PEG 20: 36 mg/m2 on Day -7 of Cycle 1, and Days 1, 8, and 15 of each 21-day cycle Gemcitabine: 600 mg/m2 on days 1 and 8 of each 21-day cycle Docetaxel: 60 mg/m2 on day 8 of each 21-day cycle
  Interventions: Drug: ADI PEG20
- PBOGemDoc (Placebo Comparator): Placebo: matched PBO on Day -7 of Cycle 1, and Days 1, 8, and 15 of each 21-day cycle Gemcitabine: 900 mg/m2 on days 1 and 8 of each 21-day cycle Docetaxel: 75 mg/m2 on day 8 of each 21-day cycle
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ADI PEG20 — Treatment for advanced or metastatic uterine/non-uterine leiomyosarcoma (LMS)
  Other Names: Pegargiminase
  Arms: ADIGemDoc
Other: Placebo — Treatment for advanced or metastatic uterine/non-uterine leiomyosarcoma (LMS)
  Arms: PBOGemDoc

SUMMARY:
To compare the efficacy and safety in subjects with advanced or metastatic LMS previously treated with an anthracycline.

DETAILED DESCRIPTION:
This is a global, multicenter, randomized, double-blind, placebo-controlled, parallel-group phase 3 trial that will compare the efficacy and safety in subjects with advanced or metastatic LMS previously treated with an anthracycline.

ELIGIBILITY:
Inclusion Criteria:

* A subject will be eligible for study participation if he/she meets the following criteria:

  1. Histologically or cytologically confirmed, grade 2 or 3, LMS STS that would be standardly treated with Gem or GemDoc.
  2. Determination of LMS subtype: uterine or non-uterine.
  3. Measurable disease per RECIST 1.1 (Appendix A), defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam.
  4. Previous treatment with up to 2 systemic regimens, including at least 1 systemic regimen containing doxorubicin.
  5. Treatment > one year ago in the adjuvant/neoadjuvant setting with Gem or Doc is allowed.
  6. Age >18 years.
  7. Eastern Cooperative Oncology Group (ECOG) performance status of < 1 at enrollment (Appendix B).
  8. Leukocytes ≥ 3,000/mcL.
  9. Absolute neutrophil count ≥ 1,500/mcL.
  10. Platelets ≥ 100,000/mcL.
  11. Hemoglobin ≥ 8.0 g/dL
  12. Total bilirubin ≤ 2 x ULN. (≤ 3 x ULN for potential subjects with Gilbert's Disease)
  13. AST(SGOT)/ALT(SGPT) ≤ 3 x ULN (or ≤ 5 x ULN if liver metastases are present)
  14. Creatinine clearance ≥ 60 mL/min (by Cockcroft-Gault equation).
  15. Serum uric acid ≤ 8 mg/dL (with or without medication control).
  16. QTc interval range from 350 to 450 ms for adult men and from 360 to 460 ms for adult women.
  17. Subjects and their partners must be asked to use appropriate contraception. They must agree to use 2 forms of contraception or agree to refrain from intercourse for the duration of the study and for 35 days after the last dose of ADI-PEG 20 or for at least 3 months (male subjects) or 6 months (female subjects) after treatment with gemcitabine, whichever is the longer duration.
  18. Ability to understand and willingness to sign the informed consent form.
  19. No concurrent investigational drug studies are allowed.

Exclusion Criteria:

* A subject will not be eligible for study participation if he/she meets any of the exclusion criteria:

  1. Subjects with history of another primary cancer, including co-existent second malignancy, with the exception of: a) curatively resected non-melanoma skin cancer; b) curatively treated cervical carcinoma in situ; or c) other primary solid tumor with no known active disease present in the opinion of the Investigator will not affect subject outcome in the setting of current diagnosis.
  2. Currently receiving chemotherapy, immunotherapy, interferon, radiation therapy or other investigational agents. Note: Chemotherapy agent washout period is 5 half-lives prior to randomization. Radiation washout period is 7 days prior to randomization.
  3. Prior treatment with ADI-PEG 20, Gem or Doc. Patients treated > one year ago in the adjuvant/neoadjuvant setting with Gem or Doc are allowed to be enrolled.
  4. Prior pelvic radiation.
  5. Known brain metastases. Such patients must be excluded from this trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
  6. History of allergic reactions attributed to compounds of similar chemical or biologic composition to ADI-PEG 20, Gem, Doc, polysorbate 80, pegylated compounds, or other agents used in this study.
  7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
  8. History of seizure disorder not related to underlying cancer.
  9. Grade 2 or higher neuropathy.
  10. Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
  11. Known HIV-positivity. Because of the potential for pharmacokinetic interactions of antiretroviral therapy with the study treatment. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
  12. Currently receiving other immunosuppressive agents.
  13. Subjects under guardianship, curatorship, under legal protection or deprived of liberty by an administrative or judicial decision

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary End Point of PFS | Subjects will receive triplet combination treatment followed by weekly monotherapy ADI-PEG 20 or PBO (Each cycle is 21 days). Subjects tolerating chemotherapy may continue chemotherapy beyond 8 cycles and up to 104 weeks (~2 years).
  The primary objective is to compare the primary endpoint of PFS in subjects treated with the arginine degrading enzyme ADI-PEG 20 plus Gem and Doc (ADIGemDoc) or PBO plus Gem and Doc (PBOGemDoc) in the 2nd or 3rd line setting using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 assessed by blinded independent central review committee (BICR)

SECONDARY OUTCOMES:
Secondary End Point of ORR (CR+PR) | Subjects will receive triplet combination treatment followed by weekly monotherapy ADI-PEG 20 or PBO (Each cycle is 21 days). Subjects tolerating chemotherapy may continue chemotherapy beyond 8 cycles and up to 104 weeks (~2 years).
  The secondary objectives are to compare ADIGemDoc versus PBOGemDoc with respect to:
  Objective response rate (ORR) (complete response [CR] + partial response [PR]) The secondary endpoint of ORR will be assessed by BICR using RECIST 1.1 and tested using a CMH test stratified by the stratification factors used during the randomization based on the ITT population.
Secondary End Point of Overall Survival (OS) | Subjects will receive triplet combination treatment followed by weekly monotherapy ADI-PEG 20 or PBO (Each cycle is 21 days). Subjects tolerating chemotherapy may continue chemotherapy beyond 8 cycles and up to 104 weeks (~2 years).
  The secondary objectives are to compare ADIGemDoc versus PBOGemDoc with respect to:
  OS
  The secondary endpoint of OS will be tested using a log-rank test stratified by the stratification factors used during the randomization based on the ITT population. A stratified Cox model will be used to estimate HR and 95% CI, and KM curves will be used to estimate OS median and 95% CI.
Secondary End Point of Safety and Tolerability | Subjects will receive triplet combination treatment followed by weekly monotherapy ADI-PEG 20 or PBO (Each cycle is 21 days). Subjects tolerating chemotherapy may continue chemotherapy beyond 8 cycles and up to 104 weeks (~2 years).
  All clinically significant abnormalities and deteriorations will be followed and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Event (NCI CTCAE V5).

CONTACTS AND LOCATIONS:
Overall Officials: John S Bomalaski, Study Director — Polaris Group
Locations (30):
- United States (25):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - USC Norris comprehensive cancer center, Los Angeles, California
  - Stanford University Medical Centre, Palo Alto, California
  - UCSF, San Francisco, California
  - UCLA, Santa Monica, California
  - University of Colorado Cancer Center/ CU Anschutz Medical Campus, Aurora, Colorado
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Miami/ Sylvester Comprehensive Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Mass General Brigham Cancer Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Wexner Medical Center/ The James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - UPenn (Abramson Cancer Center, Pennsylvania Hospital), Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin/ Froedtert Hospital, Milwaukee, Wisconsin
- Canada (2):
  - UHN - Princess Margaret Cancer Center (Ontario), Toronto, Ontario
  - McGill University Health Centre (Quebec), Montreal, Quebec
- Taiwan (3):
  - Chang Gung Medical Foundation Kaohsiung, Kaohsiung City, Niaosong District
  - National Taiwan University Hospital, Taipei, Taipei
  - Taipei Veterans General Hospital, Taipei, Taipei

IPD SHARING:
Plan to Share IPD: No